CLINICAL TRIAL: NCT01484847
Title: Pharmacokinetic Assessment of PF-00299804 in Patients With Locally Advanced Head and Neck Squamous Cell Carcinoma Following Administration Through a Gastrojejunostomy Feeding Tube
Brief Title: A Study of PF-00299804 When Given Through a Feeding Tube in Locally Advanced Head and Neck Squamous Cell Carcinoma
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Health Network, Toronto (Other)
Collaborators: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: WS1544542/Pan-HER-GT-001
Record Dates: First submitted 2011-09-30; First posted 2011-12-02 (Estimated); Last update posted 2015-07-10 (Estimated); Status verified 2015-07

CONDITIONS: Head and Neck Squamous Cell Carcinoma
Keywords: advanced; PF-00299804; head and neck; pharmacokinetic; squamous cell carcinoma; gastrojejunostomy; feeding tube
MeSH Terms: conditions — Squamous Cell Carcinoma of Head and Neck; Carcinoma, Squamous Cell | interventions — dacomitinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- PF-00299804 (Experimental): Patients with locally advanced head and neck squamous cell carcinoma will be treated with a single dose (45mg) of PF-00299804 via G-Tube on an empty stomach
  Interventions: Drug: PF-00299804

INTERVENTIONS:
Drug: PF-00299804 — Tablet, single dose of 45 mg via gastrojejunostomy tube (G-Tube) on an empty stomach

SUMMARY:
This is a study to assess how much of the investigational drug, PF-00298804, is in the blood stream over a period of time (called pharmacokinetic tests or PK) in patients with locally advanced head and neck squamous cell carcinoma who have a (gastrojejunostomy) feeding tube.

DETAILED DESCRIPTION:
This is a single arm pharmacokinetic assessment study conducted at Princess Margaret Hospital in which eligible patients will be enrolled successively to receive a single dose of PF-00299804 in an open-labelled, unblinded manner. All patients will receive 45 mg of PF-00299804 via Gastrostomy (GT) once only on an empty stomach (i.e. 2 hours before or after oral food intake or GT feeds (food intake of less than 500 calories permitted)) as an inpatient. All patients will be admitted for an overnight inpatient stay (approximately 24 hours) to facilitate pharmacokinetic assessment. There will be no dose reductions or modifications. Blood sampling for pharmacokinetics will occur on day 1 immediately prior to the dose of PF-00299804 (t=0), then at t=30 minutes, t=1 hour, t=2 hours, t=3 hours, t=4 hours, t=6 hours, t=12 hours, t=24 hours, t=48 hours, t=72 hours, t=96 hours, t=144 hours, t=168 hours, t=192 hours, and t=216 hours.

ELIGIBILITY:
Inclusion Criteria:

* Signed, voluntary informed consent provided
* Willing and able to comply with visits, treatment plan, pharmacokinetics, tests, other procedures
* Confirmed SCCHN. Other primary sites of head and neck carcinoma: nasopharynx, skin, maxillary sinus or unknown primary, are allowed
* Must have functioning gastrojejunostomy tube
* May be receiving concurrent chemoradiation, radiation alone or recently completed surgery for locally advanced disease
* Prior treatment with agents targeted to epidermal growth factor receptor not allowed.
* Any treatment-related toxicity, including laboratory abnormalities, must have recovered to CTCAE Grade 2 (v.4.0) or baseline, except toxicity not considered safety risk. Chronic dysphagia, xerostomia or other local effect from prior surgery or radiation will not be considered exclusion criterion if stable for ≥ 3 months.
* ECOG performance status 0-2
* Must have adequate organ function determined by: Serum creatinine ≤ 1.5 ULN (upper limit of normal) or calculated creatinine clearance of ≥ 50 mL/min using the formula: Creatinine clearance = [(140-age) x wt (kg) x Constant] / creatinine (µmol/L) [Constant = 1.23 for men; 1.04 for women]. Absolute neutrophil count (ANC) ≥ 1.5 x 109/L; Leukocytes ≥ 3.0 x 109/L; Hemoglobin ≥ 80 g/L (or > 8 g/dL); Platelets ≥ 100 x 109/L. Total bilirubin ≤ ULN; AST (SGOT) and ALT (SGPT) ≤ 2.5 x ULN. 12-Lead electrocardiogram (ECG) with normal tracing, or clinically non-significant with no medical intervention; QTc interval ≤ 470 msec, without history of Torsades de Pointes or other QTc abnormality

Exclusion Criteria:

* Cannot be enrolled on another clinical trial
* Prior investigational drug therapy within 30 days or 5 half-lives preceding first dose of study drug (whichever longer)
* Requirement for drugs highly dependent on CYP2D6 for metabolism since PF-00299804 is a potent CYP2D6 inhibitor
* Patients currently taking drugs with risk of Torsades de Pointes
* Any acute/chronic medical, psychiatric condition or laboratory abnormality that could increase risk of participation, trial drug administration or interfere with interpretation of trial results and, investigator feels, would make patient inappropriate for entry. Including: History of interstitial lung disease; Uncontrolled hypertension, unstable angina, myocardial infarction, symptomatic congestive heart failure within past year, uncontrolled cardiac arrhythmia, diagnosed/suspected congenital long QT syndrome; history of stroke, deep vein thrombosis, or stable for 6 months without requiring antiarrhythmics/significant change in medical management; Active bacterial, fungal or viral infection including hepatitis B/C, and human immunodeficiency virus. Testing not required at baseline with no symptoms of infection. History of significant bleeding disorder, or concurrent medications that investigator feels may lead to unacceptable coagulation during perioperative interval, including: congenital bleeding disorders; acquired bleeding disorder within a year
* Other serious uncontrolled medical disorder or active infection that would impair ability to receive study treatment as determined by investigator
* Dementia or altered mental status that would limit ability to obtain informed consent and compliance with requirements of the protocol
* Patients breastfeeding or pregnant are excluded. Those with reproductive potential must have negative pregnancy test within 72 hours of treatment. Patients of reproductive potential include any female who has experienced menarche and who has not undergone successful surgical sterilization, or is not postmenopausal. Patients of reproductive potential/partners must agree to effective contraception while receiving trial treatment and for at least 3 months after. Effective contraception will be judgment of principal investigator or designate
* Inability/lack of willingness to comply with visits, treatment plans, assessments or tests

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2011-12; Primary Completion 2013-03 (Actual); Study Completion 2015-07 (Actual)

PRIMARY OUTCOMES:
Composite (or Profile) of Pharmacokinetics Time Frame: predose, 0,1,2,3,4,6,8,12,24,48,72, 96 hours post-dose | 3-6 months
  Cmax, Area Under Curve, Tmax

SECONDARY OUTCOMES:
Comparison of pharmacokinetic parameters of study subjects with existing phase I pharmacokinetic data following administration of PF-00299804. | 3-6 months
  Tmax=4-24 hrs, Cmax = 28.1 ng/ml, AUCtau=47 hr*ng/ml, t1/2=85.1
Overall safety profile as per National Cancer Institute Common Terminology Criteria for Adverse Events version 4.0. | 3-6 months

CONTACTS AND LOCATIONS:
Overall Officials: Lillian Siu, MD, Principal Investigator — University Health Network/Princess Margaret Hospital
Locations (1):
- Princess Margaret Hospital, Toronto, Ontario, Canada